CLINICAL TRIAL: NCT06245850
Title: Impact of Baduanjin Exercise Combined With Rational Emotive Behavior Therapy on Sleep and Mood in Patients With Post-stroke Depression: A Randomized Controlled Trial
Brief Title: Impact of Baduanjin Exercise Combined With Rational Emotive Behavior Therapy on Sleep and Mood in Patients With Post-stroke Depression
Acronym: ZZU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Liu Yihan, resident doctor, Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zhengzhouuniversity; 82071331 (Other Grant/Funding Number: National Natural Science fouding)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin Group (Experimental)
  Interventions: Behavioral: Baduanjin
- REBTgroup (Active Comparator)
  Interventions: Behavioral: Rational emotive behavior therapy

INTERVENTIONS:
Behavioral: Baduanjin — chinese baduanjin
  Arms: Baduanjin Group
Behavioral: Rational emotive behavior therapy — Rational emotive behavior therapy
  Arms: REBTgroup

SUMMARY:
Patients and their families all agreed .

ELIGIBILITY:
Inclusion Criteria:

1. Conformity to the diagnostic criteria for stroke in the "Diagnostic Essentials of Various Cerebrovascular Diseases" revised by the Fourth National Cerebrovascular Academic Conference, and confirmed by cranial CT or MRI.
2. The course of stroke was 2 weeks to 6 months, with steady conditions and stable vital signs.
3. The age ranged from 30 to 80 years old, with at least a junior high school education.
4. The patients had no serious intellectual, language comprehension and behavioral disorders, and could complete the assessment of scales.
5. Achieving a sitting balance of at least reaches level 3, Brunnstrom stage IV or above, and being able to complete Baduanjin training.
6. The National Institutes of Health Stroke Scale (NIHSS) ≤ 15 points.
7. Conforming to the diagnostic criteria for depression in the "Chinese Experts Consensus on Clinical Practice of Post-Stroke Depression".

Exclusion Criteria:

The exclusion criteria:

1. Disturbance of consciousness, unable to cooperate with polysomnography (PSG) and scale evaluators.
2. Pre-existing diagnosis of depression before stroke.
3. Severe pre-existing sleep disorders before stroke.
4. Patients with mental illness, immune system disorders, severe liver and kidney dysfunction, and severe cardiopulmonary dysfunction

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
HAMD score | 8 weeks
  HAMD score: The Hamilton Depression Scale (HAMD) were used to evaluate the depression level of the subjects. The HAMD-17 score is 0-6 points for no depression, 8 7-17 points for mild depression, 18-24 points for moderate depression, and 25-54 points for severe depression. A higher score corresponds to more severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No